CLINICAL TRIAL: NCT02863146
Title: Efficacy of the Use of a Refrigerant Helmet to Prevent Alopecia in Patients Treated With Eribulin for Locally Advanced or Metastatic Breast Cancer Pretreated With Anthracyclines and Taxanes
Brief Title: Efficacy of the Use of Refrigerant Helmet to Prevent Alopecia in Patients Treated With Eribulin for Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HALACAP-1406
Record Dates: First submitted 2016-02-15; First posted 2016-08-11 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: locally advanced breast cancer; alopecia; eribulin
MeSH Terms: conditions — Breast Neoplasms; Alopecia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
HALACAP-1406 is a prospective single-centre non-interventional study assessing the refrigerant helmet use as medical device to prevent alopecia induced by eribulin (Halaven®) in the conditions of use specified in its marketing authorization. Eribulin will be used alone for the treatment of the patients having a locally advanced or metastatic breast cancer which have progressed after at least 1 chemotherapy regimen for their advanced stage.

DETAILED DESCRIPTION:
A nurse will meet the patient and present the study, then the patient will be invited to participate. If the patient is interested, an information note will be given and the non-opposition of the patient will be collected.

Patients will be registered via a registration form and an inclusion number will be attributed at each patient.

Eribulin will be used within the framework of its marketing authorization, per cycle of 21 days, at day 1 and day 8.

Modalities of refrigerant helmet use will be set according to the habits of the Oscar Lambret center with the following rules :

* Placement of a single-use non-woven hygiene cap on the scalp
* T-15 minutes: placement of the refrigerant helmet
* T0: begin of eribulin infusion (duration: 2-5 minutes)
* T+15 minutes: rinse of the line
* T+30 minutes: withdrawal of the helmet

Efficacy will be evaluated before treatment and at each eribulin cycle.

ELIGIBILITY:
Inclusion Criteria:

* Female patient who has a locally advanced or metastatic breast cancer
* Indication of Halaven treatment :

patient pretreated with anthracyclines or taxanes, patient who has received at least 1 chemotherapy regimen for their advanced or metastatic stage

* Patient who has had enough time to have retrieved her hair or whose last chemotherapy regimen didn't induce alopecia.
* Aged ≥ 18 years
* Non-opposition of the patient must have been collected

Exclusion Criteria:

* Skin metastasis of the scalp
* Sensitivity to cold, cold agglutinin disease or cryoglobulinemia
* Impossibility to submit at the study procedures due to geographic, social or mental reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic breast cancer patients treated with eribulin and whose cancer has progressed after at least 1 chemotherapy regimen for their advanced stage
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Alopecia grade after 3 cycles of eribulin according to NCI-CTCAE v4.0 | on the day 1 of cycle 4
  Efficacy of the refrigerant helmet : Alopecia grade after 3 cycles of eribulin

SECONDARY OUTCOMES:
Adverse events graded according to NCI-CTCAE v4.0 | every 28 days : at day 1 of each cycle during 3 cycles
  Tolerance of the refrigerant helmet : graduation of adverse events lived by patients

CONTACTS AND LOCATIONS:
Overall Officials: Laurence VANLEMMENS, MD, Principal Investigator — Centre Oscar Lambret; Monique Blondel, Study Director — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No